CLINICAL TRIAL: NCT00777062
Title: A Phase II, Randomized, Double-Blind Pilot Trial of VIVITROL® (Naltrexone for Extended-Release Injectable Suspension) for the Treatment of Cocaine and Alcohol Dependence
Brief Title: VIVITROL as a Treatment for Cocaine and Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Alkermes, Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kyle Kampman, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 808641; 5P50DA012756-10 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Cocaine Dependence; Alcohol Dependence
Keywords: alcohol; cocaine; addiction; alcoholism; substance dependence; substance abuse
MeSH Terms: conditions — Cocaine-Related Disorders; Alcoholism; Behavior, Addictive; Substance-Related Disorders | interventions — vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): VIVITROL (Naltrexone extended-release injectable suspension), 380 mg injection at the start of weeks 2 and 6
  Interventions: Drug: VIVITROL (Naltrexone extended-release injectable suspension)
- 2 (Placebo Comparator): Placebo injection, 380 mg injection at the start of weeks 2 and 6.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIVITROL (Naltrexone extended-release injectable suspension) — VIVITROL (Naltrexone extended-release injectable suspension), 380 mg injection at the start of weeks 2 and 6.
  Other Names: Vivitrol
  Arms: 1
Drug: Placebo — Placebo injection at the start of weeks 2 and 6.
  Arms: 2

SUMMARY:
To evaluate the efficacy of VIVITROL (naltrexone for extended-release injectable suspension) for the treatment of co-occurring cocaine and alcohol dependence

DETAILED DESCRIPTION:
This is a Phase II double-blind randomized controlled clinical pilot study. The exploratory objectives in the proposed study will be examined with a 2-group design to assess the efficacy of naltrexone extended-release injectable suspension (VIVITROL™) as compared to placebo. Safety measures will be collected weekly through medical management (MM) by medical practitioners, including adverse events and concomitant meds. The psychosocial treatment will be Cognitive Behavioral Coping Skills Therapy (CBT). Subjects will be 80 men and women with current DSM-IV diagnoses of alcohol dependence and cocaine dependence that will be randomized to receive either VIVITROL or placebo (40 subjects per group). All subjects will receive weekly sessions of CBT and MM. The study length for each subject is comprised of 1-3 weeks of screening, an 8-week double-blind, placebo-controlled trial with MM and CBT (medication phase), and an end of medication visit.

Primary Exploratory Objectives:

* To compare medication groups' rates of cocaine abstinence, as determined by urine assay for benzoylecgonine (BE), the primary metabolite of cocaine. This will be cross-checked against participants' self-reports of cocaine use through Time-Line Follow Back (TLFB)(Sobell & Sobell, 1992).
* To compare medication groups' rates of abstinence from drinking, and of clinically significant drinking, as measured by the TLFB.

Secondary Exploratory Objectives:

* To evaluate medication groups' reports of craving for cocaine and alcohol, as measured by scores on the Penn Alcohol Craving Scale and the Minnesota Cocaine Craving Scale during the medication treatment phase.
* To compare women's reports of medication tolerance of naltrexone extended-release injectable suspension versus high dose oral naltrexone that was reported in our recently published pilot trial of high dose naltrexone for dual cocaine and alcohol dependence (Pettinati et al., 2008).

ELIGIBILITY:
Inclusion Criteria

1. Males and females, 18 to 65 years old.
2. Meets DSM-IV criteria for Cocaine Dependence, as determined by the Structured Clinical Interview for DSM-IV (SCID).
3. Meets DSM-IV criteria for Alcohol Dependence, as determined by the Structured Clinical Interview for DSM-IV (SCID).
4. Meets the following drinking criteria as measured by the Timeline Followback (TLFB) (Sobell, 1995)

   1. drank within 30 days of intake day,
   2. reports a minimum of XX standard alcoholic drinks in a consecutive 30-day period over the 90-day period prior to starting intake, and
   3. has 2 or more days of heavy drinking
5. In the past 30 days prior to consent, used no less than $ of cocaine.
6. Live within a commutable distance of the Treatment Research Center (TRC) at the Penn/VA Center for Studies of Addiction, University of Pennsylvania. We define this to be a distance within the service area of Septa, within an hour drive, or a distance that both the patient and Principal Investigator (PI) find acceptable.
7. Understands and signs the informed consent.
8. Three consecutive days of abstinence from alcohol, and a Clinical Institute Withdrawal Scale for Alcohol (CIWA-AR) (Sullivan, 1989) score below eight.

4.2 Exclusion Criteria:

1. Positive urine drug screen and/or current DSM-IV diagnosis of any psychoactive substance dependence other than cocaine, alcohol, or nicotine dependence, as determined by the SCID.
2. Concomitant treatment with psychotropic medications, including opioid analgesics.
3. Patients mandated to treatment based upon a legal decision or as a condition of employment.
4. Current severe psychiatric symptoms, e.g., psychosis, dementia, suicidal or homicidal ideation, mania or depression requiring antidepressant therapy in the opinion of the Principal Investigator (PI).
5. Taken any investigational medication within the past 30 days.
6. History within the six months prior to randomization of significant heart disease (an arrhythmia which required medication, Wolff-Parkinson-White Syndrome, angina pectoris, documented history of myocardial infarction, heart failure). These are to be reviewed on a case-by-case basis: EKG 1st degree heart block, sinus tachycardia, left axis deviation, and nonspecific ST or T wave changes are allowed; liver function tests [LFTs] <3 x ULN are acceptable).
7. Known hypersensitivity to naltrexone, PLG, carboxymethylcellulose, or any other components of the diluent.
8. Subjects with a BMI of 40 and above, as determined by the Body Mass Index Table, or that have distribution of adipose tissue such that they would be at greater risk of serious injection site reaction, based on clinical judgment. Participants with a BMI over 30 will have additional screening procedures conducted to determine inclusion in the study. These procedures include an additional screening measurement of waist-hip ratio for those participants with a BMI over 30. Males with a waist to hip ratio of >0.9 and females with a waist to hip ratio of >0.85 will be referred to the investigator for final decision of study inclusion. If the ratio is <0.9 for men or <0.85 for women they will be eligible for study inclusion without further action.
9. Patients with any serious illnesses that may require hospitalization during the study.
10. Female subjects who are pregnant or lactating, or female subjects of child-bearing potential who are not using acceptable methods of birth control. Acceptable methods of birth control include:
11. Clinical laboratory tests (CBC, blood chemistries, urinalysis) outside normal limits that are clinically unacceptable to the Principal Investigator.
12. Current physiological opioid dependence.
13. Experiencing acute opiate withdrawal.
14. Likely to receive scheduled surgery, which may require treatment with opioid analgesics.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Pettinati, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: University of Pennsylvania Center for the Studies of Addiction — http://www.med.upenn.edu/csa/index.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Vivitrol: VIVITROL (Naltrexone extended-release injectable suspension), 380 mg injection at the start of weeks 2 and 6
- Placebo: Placebo injection, 380 mg injection at the start of weeks 2 and 6.
Period: Overall Study
Arm/Group | Vivitrol | Placebo
Started | 39 | 41
Completed | 36 | 36
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vivitrol | Placebo | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 41 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (7.0) | 48.4 (6.3) | 47.9 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 30 | 35 | 65
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: Urine Assay for Benzoylecgonine (BE), the Primary Metabolite of Cocaine.
Description: Percentage of subjects with no cocaine use for at least 3 weeks
Time Frame: 8 week medication phase
Measure: Number; unit: Percentage of Participants
Arm/Group | Vivitrol | Placebo
Number analyzed (Participants) | 39 | 41
Percentage of Participants | 33.3 | 31.7

2. Primary Outcome: Time Line Follow Back -Reported Days of Abstinence From Drinking
Description: Percentage of participants who were abstinent from drinking
Time Frame: 8 week medication phase
Measure: Number; unit: Percentage of Participants
Arm/Group | Vivitrol | Placebo
Number analyzed (Participants) | 39 | 41
Percentage of Participants | 10.3 | 17.1

ADVERSE EVENTS:
Arm/Group | Vivitrol | Placebo
Serious Adverse Events (participants affected / at risk) | 5/39 | 4/41
Other Adverse Events (participants affected / at risk) | 22/39 | 13/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivitrol (N=39) | Placebo (N=41)
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Participant sent to dermatology clinic and they recommended monitoring the site, but no urgent action needed. Participant t finished out study visits and swelling went down.
Hospitalization for Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Hospitalization for pneumonia (General disorders) | 0 (0) | 1 (1) — Participant complained of feeling ill and very fatigued. He had a high fever on 8/5/11, so study nurse recommended that he go to the ER. He was admitted on 8/5/11 with pneumonia, and released on 8/9/11.
Worsening of addiction symptoms (General disorders) | 1 (1) | 1 (1) — Participant entered inpatient treatment for worsening of addiction symptoms.
Lacerations and fractured rib (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Participant was physically attacked and hospitalized for injuries.
Hospitalization for nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant said nausea was resolved on 3/7/10 and did not receive second injection. He finished his final study visit on 4/12/10.
Hospitalization for an overdose of tylenol (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vivitrol (N=39) | Placebo (N=41)
Swelling at the injection site (Skin and subcutaneous tissue disorders) | 22 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No